CLINICAL TRIAL: NCT07032909
Title: Evaluating the Effectiveness of Comfort Reading Mode in Preventing Dry Eyes and Visual Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TREC2025-KY099
Record Dates: First submitted 2025-05-20; First posted 2025-06-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Visual Fatigue
Keywords: electronic display; visual fatigue; tear break-up time; visual function; critical flicker fusion frequency
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Intervention Model Description: This study is designed with a total of five groups, where participants will sequentially and randomly undergo all the intervention procedures.
Who Masked: Investigator
Masking Description: In order to eliminate the influence of subjective factors during the examination, this study was blinded only to the examiner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- yellow background and black text mode 1 Group (Experimental): This is the group that performs visual evoked tasks using yellow background and black text mode 1. In this group, the impact of the same text content on the visual fatigue, and tear break-up time were assessed, including but not limited to indicators such as reading efficiency, blinking detection, visual function and retinal fundus blood flow.
  Interventions: Behavioral: comfortable reading mode
- yellow background and black text mode 2 Group (Experimental): This is the group that performs visual evoked tasks using yellow background and black text mode 2. In this group, the impact of the same text content on the visual fatigue, and tear break-up time were assessed, including but not limited to indicators such as reading efficiency, blinking detection, visual function and retinal fundus blood flow.
  Interventions: Behavioral: comfortable reading mode
- black background and white text mode Group (Experimental): This is the group that performs visual evoked tasks using black background and white text mode. In this group, the impact of the same text content on the visual fatigue, and tear break-up time were assessed, including but not limited to indicators such as reading efficiency, blinking detection, visual function and retinal fundus blood flow.
  Interventions: Behavioral: comfortable reading mode
- black background and yellow text mode Group (Experimental): This is the group that performs visual evoked tasks using black background and yellow text mode. In this group, the impact of the same text content on the visual fatigue, and tear break-up time were assessed, including but not limited to indicators such as reading efficiency, blinking detection, visual function and retinal fundus blood flow.
  Interventions: Behavioral: comfortable reading mode
- white background and black text mode Group (No Intervention): This is the group that performs visual evoked tasks using white background and black text mode. In this group, the impact of the same text content on the visual fatigue, and tear break-up time were assessed, including but not limited to indicators such as reading efficiency, blinking detection, visual function and retinal fundus blood flow.

INTERVENTIONS:
Behavioral: comfortable reading mode — Subjects are asked to read a terminal display device for 45 minutes, featuring texts with different reading mode treatments. Specifically, they will read the same text content for 45 minutes with different background and text color. The participants will complete a total of 4 sets of tests in a random order.
  Arms: black background and white text mode Group; black background and yellow text mode Group; yellow background and black text mode 1 Group; yellow background and black text mode 2 Group

SUMMARY:
The purpose of this study was to investigate the effects of visual fatigue and dry eye level under different reading background polarities and different text colours, and to evaluate the effect of comfortable reading mode on the improvement of visual fatigue and dry eye level

DETAILED DESCRIPTION:
The effect of electronic display devices on visual fatigue of human eyes was the primary evaluation index and the primary outcome index of this experiment. Secondary outcome indicators were tear film break-up time, tear film height, and subjective visual fatigue score. Other outcome indicators were blink detection, ocular axial length measurement, accommodative function and retinal fundus blood flow. Baseline values of the above metrics were measured separately before each group of trials and then, after 45 minutes of e-text reading, specific values of the different metrics were collected when using different reading modes and all valid measurements were statistically compared and analysed. To assess the effect of comfortable reading modes on reducing visual fatigue and dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult population, regardless of gender.
* Refractive error is less than or equal to -2.5D and both eyes achievecorrected visual acuity of 0.8 or higher.
* Normal intraocular pressure with no organic pathology.
* No apparent symptoms of dry eye.
* Willing to cooperate to complete all the tests.
* Voluntarily signing the informed consent form.

Exclusion Criteria:

* Individuals with strabismus and amblyopia exist.
* Suffering from congenital eye conditions such as congenital cataracts or congenital retinal diseases.
* Those who have undergone intraocular surgery (such as cataract removal, intraocular lens implantation, etc.).
* Individuals with refractive media opacity (such as corneal lesions, lens opacity, etc.).
* Only one eye meets the inclusion criteria.
* Active corneal infections such as bacterial, fungal, viral, or other acute or chronic anterior segment inflammations.
* Currently using medications that may lead to dry eye or affect vision and corneal curvature.
* Other ocular conditions, such as dacryocystitis, eyelid disorders and abnormalities, abnormal intraocular pressure, and glaucoma.
* Unable to undergo regular eye examinations.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Critical flicker fusion frequency | Participants underwent five randomized experimental conditions through study completion, an average of 2 months. For each condition, CFF test was administered at baseline (pre-experiment) and post-task,totaling ten completions per participant.
  Critical flicker fusion frequency was measured before and after the task by a flicker fusion frequency detection device to assess changes in the degree of ocular fatigue. To compare the difference in CFF after wearing anti-blue glasses with normal glasses and to evaluate the effect of anti-blue glasses in preventing asthenopia.

SECONDARY OUTCOMES:
Visual fatigue | Participants underwent five randomized experimental conditions through study completion, an average of 2 months. For each condition, visual fatigue test was administered at baseline and post-task,totaling ten completions per participant.
  The visual fatigue questionnaire utilized in this study consists of a self-report survey with a total of 19 items. It is designed to comprehensively assess the severity of visual fatigue symptoms, with a scoring system ranging from 1 to 7. Higher scores indicate more severe symptoms, encompassing three primary domains: ocular symptoms, visual discomfort, and psychological aspects triggered by visual fatigue.
Break up time | Participants underwent five randomized experimental conditions through study completion, an average of 2 months. For each condition, BUT test was administered at baseline and post-task,totaling ten completions per participant.
  This clinical study included tear film breakup time measurement using fluorescein sodium stained paper immediately after each VDT task, reflecting tear film stability, and evaluating the degree of dry eye
Measurement of Accommodative Sensitivity with Flip-Chart Post-VDT Tasks | Participants underwent five randomized experimental conditions through study completion, an average of 2 months. For each condition, AC/A test was administered at baseline and post-task,totaling ten completions per participant.
  This clinical study involves the assessment of accommodative sensitivity for both monocular and binocular vision using a flip-chart immediately following each VDT task. The measurement will quantify the number of optotypes correctly identified within one minute, indicative of the subject's accommodative capacity.
equivalent refraction | Participants underwent five randomized experimental conditions through study completion, an average of 2 months. For each condition, SE test was administered at baseline and post-task,totaling ten completions per participant.
  This clinical study included testing subjects for equivalent refraction diopters, which can indirectly reflect changes in the degree of myopia in the eye after the use of VDT at close range

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University,, Beijing, Beijing/China, China

IPD SHARING:
Plan to Share IPD: No